CLINICAL TRIAL: NCT07126522
Title: Advancing Survivorship Support Through Virtual Health Equity Resources for Breast Cancer Responsive Education (HERCaRE)
Brief Title: Virtual Support Platform (HERCaRE Application) for the Improvement of Survivorship Among Black Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-001524; NCI-2025-05318 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 25-001524 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (HERCaRE app) (Experimental): Patients use the HERCaRE app over 4-6 weeks on study.
  Interventions: Other: Discussion; Other: Internet-Based Intervention; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Discussion — Ancillary studies
  Other Names: Discuss
Other: Internet-Based Intervention — Use the HERCaRE app
Other: Interview — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well a virtual support platform, the Health Equity Resources for Breast Cancer Responsive Education (HERCaRE) application (app), works in improving survivorship among Black survivors of breast cancer. The HERCaRE platform is a mobile-friendly app that includes culturally tailored educational materials, interactive content, and health equity resources to help patients better understand and manage survivorship after breast cancer treatment. This trial may help improve how digital health interventions can enhance survivorship support and access to resources.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Self-identified Black women with a history of breast cancer

  * "Self-identified Black woman" refers to individuals who personally identify as a Black or African American woman, inclusive of cisgender women from diverse cultural backgrounds. This will be confirmed during a verbal eligibility screening conducted prior to enrollment
* Completed active breast cancer treatment (e.g., surgery, chemotherapy, or radiation) at least one month prior to enrollment; survivors receiving long-term hormonal therapy are also eligible
* Reside within the Mayo Clinic Florida catchment area
* Have access to a smartphone or willingness to use alternative access points

  * "Alternative access points" refer to non-clinical settings through which participants may be made aware of the study, including support groups, community health events, churches, and partner organizations that engage with breast cancer survivors outside of the traditional healthcare setting

Exclusion Criteria:

* Individuals without a history of breast cancer
* Those unable to provide verbal consent
* Individuals who lack the ability to engage with digital platforms, as determined during the screening process via brief questions assessing comfort and experience with mobile technology. Participants must be able to open the app, read content, and complete survey independently. iPads will be available for participants who do not have their own mobile device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Survivorship engagement - login | Up to 6 weeks
  Assessed by active use of the Health Equity Resources for Breast Cancer Responsive Education (HERCaRE) platform, defined as number of logins per participant.
Survivorship engagement - time | Up to 6 weeks
  Assessed by the length of time each participant spent using the HERCaRE platform.
Survivorship engagement - self-report | Up to 6 weeks
  Assessed by self-reported actions such as initiating conversations with providers or accessing survivorship resources. Information will be obtained through semi-structured interviews.
Adherence to follow-up care | Up to 6 weeks
  Assessed by participant self-reported scheduling or completion of appointments (e.g., mammograms, primary care physician visits). Information will be obtained through semi-structured interviews.

SECONDARY OUTCOMES:
Participant satisfaction - HERCaRE Final Survey | Up to 6 weeks
  Will be assessed by 5 question from a 9-question HERCaRE Final Survey. Three questions are answered on a 5-point scale (strongly agree, agree, neutral, disagree, strongly disagree), and two questions are open-ended/free text.
Perceived usability - HERCaRE Final Survey | Up to 6 weeks
  Will be assessed by a 4 question of a 9-question HERCaRE Final Survey. Two questions are multiple choice (e.g., Yes, No, Not sure) Once is related to likelihood of taking follow-up actions such as "schedule and attend a follow-up appointment" or "ask more questions during my next visit." The final question is an open-ended/free text question related to any difficulties using the app or competing activities.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Salinas, DrPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials